CLINICAL TRIAL: NCT04896879
Title: Rectal Cancer Survivorship, the Struggle of the Low Anterior Resection Syndrome (LARS). Experiences and Needs of Patients, Their Informal Caregiver and Healthcare Professionals
Brief Title: Experiences and Needs of Patients, Their Informal Caregiver and Healthcare Professionals Regarding LARS
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Kom Op Tegen Kanker (Other); AZ Sint-Jan AV (Other); AZ Delta (Other); AZ Sint-Lucas Gent (Other)
Responsible Party: Principal Investigator, GIHeelkunde, Principal investigator, University Hospital, Ghent
Other Study IDs: EC2016/1016
Record Dates: First submitted 2020-12-31; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Low Anterior Resection Syndrome; Rectal Cancer
Keywords: low anterior resection syndrome
MeSH Terms: conditions — Low Anterior Resection Syndrome; Rectal Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients: Patients with major LARS
  Interventions: Behavioral: interviews
- Informal caregivers: Informal caregivers of patients with major LARS
  Interventions: Behavioral: interviews
- Healthcare professionals: Healthcare professionals taking care for patients with LARS
  Interventions: Behavioral: interviews

INTERVENTIONS:
Behavioral: interviews — semi-structured interviews will be conducted in patients with major LARS and their informal caregiver to explore their experiences and needs. Focus groups will be perfomed with healthcare professionals of several professions.

SUMMARY:
Exploration of the experiences and needs of patients with the low anterior resection syndrome, their informal caregiver and health care professionals. This is a qualitative study where semi-structured interviews will be conducted with patients and informal caregivers. next to that focus groups will be performed with healthcare professionals from different professions.

ELIGIBILITY:
PATIENTS

Inclusion Criteria:

* adult patients (18+)
* confronted with major low anterior resection syndrome after rectal cancer surgery

Exclusion Criteria:

* stoma at time interview
* abdominal perineal resection

INFORMAL CAREGIVERS Inclusion criteria

* Adults (18+)
* Nominated by the participating patient as their principal caregiver Exclusion criteria None

HEALTHCARE PROFESSIONALS inclusion criteria

* Adults (18+)
* Caring for patients with LARS Exclusion criteria None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be patients with major LARS, their informal caregivers and healthcare professionals
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2016-11-22 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
needs and experiences of patients with major lars and their informal caregiver through individual semistructered interviews | Interview will last about 60 minutes
  Exploring needs and experiences of patients with major lars and their informal caregiver through individual semistructured interviews
Needs and experiences of healthcare professionals caring for patients with LARS through focus groups | Focus group will last about 60 minutes
  Exploring needs and experiences of healthcare professionals caring for patients with LARS

REFERENCES:
- [Derived] Pape E, Decoene E, Debrauwere M, Van Nieuwenhove Y, Pattyn P, Feryn T, Pattyn PRL, Verhaeghe S, Van Hecke A; Belgian LARS collaborative group. Information and counselling needs of patients with major low anterior resection syndrome: A qualitative study. J Clin Nurs. 2023 Apr;32(7-8):1240-1250. doi: 10.1111/jocn.16277. Epub 2022 Mar 6. PMID 35253296